CLINICAL TRIAL: NCT04133311
Title: A Phase III, Multinational, Multicenter, Investigator-Masked, Randomized, Active Controlled Trial, Comparing the Efficacy and Safety of DE-130A With Xalatan® in Patients With Open-Angle Glaucoma or Ocular Hypertension Over a 3-Month Period, Followed by a 12-Month Follow-Up With Open-Label DE-130A Treatment.
Brief Title: A Phase III Multinational Multicenter Investigator-Masked Randomized Active-Controlled Trial Comparing the Efficacy and Safety of DE-130A With Xalatan® in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0130A01SA
Record Dates: First submitted 2019-10-04; First posted 2019-10-21 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Open-Angle Glaucoma or Ocular Hypertension; Ocular Surface Disease
Keywords: IOP; OSD
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DE-130A (Experimental): Instillation of one drop, once daily in the evening (9 pm ±1 hour) in the conjunctival sac of the affected eye(s). Both eyes will be treated unless the patient suffers from unilateral OAG/OHT
  Interventions: Drug: DE-130A
- Xalatan® (Active Comparator): Instillation of one drop, once daily in the evening (9 pm ± 1 hour) in the conjunctival sac of the affected eye(s). Both eyes will be treated unless the patient suffers from unilateral OAG/OHT
  Interventions: Drug: Xalatan®
- DE-130A/DE-130A (Other): After 12 weeks, continue to use DE-130A once daily for an additional 12 months.
  Interventions: Drug: DE-130A/DE-130A
- Xalatan®/DE-130A (Other): After 12 weeks, use DE-130A instead of Xalatan® once daily for an additional 12 months.
  Interventions: Drug: Xalatan®/DE-130A

INTERVENTIONS:
Drug: DE-130A — Latanoprost 50 microg/ml eye drops emulsion, preservative-free eye drops emulsion in single-dose containers.
  Other Names: Catiolanze®
  Arms: DE-130A
Drug: Xalatan® — Latanoprost 50 microg/ml eye drops solution, eye drops in 2.5 ml dropper containers.
  Arms: Xalatan®
Drug: DE-130A/DE-130A — After Week 12, received DE-130A continuously.
  Other Names: Catiolanze®
  Arms: DE-130A/DE-130A
Drug: Xalatan®/DE-130A — From week 12 onwards, DE-130A was continued to be administered instead of Xalatan®.
  Other Names: Catiolanze®
  Arms: Xalatan®/DE-130A

SUMMARY:
A Phase III, Multinational, Multicenter, Investigator-Masked, Randomized, Active-Controlled Trial, comparing the efficacy and safety of DE-130A with Xalatan® in Patients with Open-Angle Glaucoma or Ocular Hypertension over a 3-Month period, followed by a 12-Month Follow-Up with Open-Label DE-130A Treatment.

DETAILED DESCRIPTION:
Phase III, prospective, interventional, multinational, multicentre, investigator-masked, randomized, active-controlled trial

Study duration:

* 5 days to 5-week washout period
* 15 months for the first 130 patients
* 12 weeks for the next 250 patients

Patients will attend 6 visits following the wash-out phase (up to 5 weeks):

* Period 1 (3-month investigator-masked treatment period, DE-130A vs Xalatan®): Randomization/Baseline visit (Day 1), Week 4 (±3 days) and Week 12 (±3 days)
* Period 2 (12-month follow-up from Week 12, open-label DE-130A treatment for the first 130 patients who complete their week 12 visit and agree to participate in the open-label period of the study): Month 6 (± 7days), Month 9 (±7 days) and Month 15 (± 1 week) visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older
2. The patient has signed and dated a written informed consent form and any required privacy authorization prior to the conduct of any study procedures.
3. Diagnosis of OAG (primary open angle glaucoma, pseudo exfoliative glaucoma, or pigmentary glaucoma), or OHT in eligible eye(s) currently on monotherapy.
4. Unilateral OAG, or OHT are permissible as long as the physician does not anticipate significant IOP changes to the fellow eye that would require treatment during the duration of the study.
5. Current treatment with monotherapy for OAG or OHT with a controlled IOP ≤ 18 mmHg in each eye (pre-washout).
6. Stable visual field (based on at least two visual fields available within the last 18 months prior to screening, including one in the last 6 months; A visual field test will be performed at screening if not already performed within the last 6 months prior to screening) in each eye.
7. Post-washout IOP ≥ 22 mmHg in at least one eye (defined at baseline visit [Day 1] by IOP measurement at both 9:00 am ± 1 hour and 4:00 pm ±1 hour)
8. Post-washout IOP ≤ 32 mmHg (defined at baseline visit [Day 1] by IOP measurement at both 9:00 am ±1 hour and 4:00 pm ±1 hour) in both eyes.
9. Ability to discontinue their current topical IOP-lowering medication for the required washout period. Washout periods should be as follows;

   * Prostaglandin analogs = 4 weeks
   * Topical beta blockers ≥ 3 weeks and ≤ 4 weeks
   * Topical carbonic anhydrase inhibitors ≥ 5 days and ≤ 4 weeks
   * All other IOP lowering medication ≥ 2 weeks and ≤ 4 weeks
10. Snellen best corrected visual acuity score of 20/100 or better in each eye
11. Patient must be willing to discontinue wearing contact lenses during the study.
12. Adequate health for study participation as determined by the investigator
13. In the opinion of the investigator, the patient is capable of understanding and complying with protocol requirements
14. Patient must be willing and able to undergo and return for scheduled study-related examinations.

    -

Exclusion Criteria:

1. Any form of glaucoma other than primary open angle glaucoma, pseudo exfoliative glaucoma, and pigmentary glaucoma in either eye.
2. IOP at any time point during the Screening or Baseline visits (Visits 1 or 2) of > 32 mmHg in either eye.
3. Current treatment for glaucoma with a fixed-combination therapy or more than one drug in either eye or with an oral drug within 6 months prior to screening.
4. Corneal abnormalities that would interfere with accurate IOP readings with an applanation tonometer in either eye.
5. Central corneal thickness ≤ 480 µm or ≥ 600 µm in either eye (historical data or at the screening visit).
6. Significant visual field loss (absolute defect in the 10° central point or mean deviation worse than -12 dB) or progressive field loss during the year before screening in either.
7. Significant optic nerve abnormality, other than glaucomatous abnormalities in the opinion of the investigator as determined by ophthalmoscopy in either eye.
8. Significant changes of the optic neuropathy (e.g. increase cupping since the last examination, optic nerve hemorrhage) in either eye.
9. Inability to visualize the patient's optic nerve in either eye.
10. Gonioscopy consistent with potential angle closure glaucoma in either eye.
11. Patients with severe blepharitis and/or Meibomian Gland Disease (MGD). Patients enrolled with mild to moderate blepharitis and/or MGD should be treated as appropriate during the study in either eye.
12. Use of oral or topical ophthalmic steroid within the past 14 days from screening date, or anticipated need for ocular steroid treatment during the study in either eye.
13. Use of intravitreal or peribulbar injection of depot steroid or placement of an intravitreal steroid implant within the past 3 months from screening date in either eye.
14. Known allergy or sensitivity to the study medications.
15. Active or expected ocular allergy during period 1.
16. Any active ocular disease (e.g. uveitis, ocular infection, severe dry eye with CFS grade 4 or more on the modified Oxford scale) in either eye. Patients may have mild cataracts, age-related maculopathy or background diabetic retinopathy if, in the opinion of the Investigator, it would not interfere with the conduct of the study.
17. Intraocular surgery within 6 months prior to screening in either eye.
18. Past history of any filtering surgery for glaucoma in either eye.
19. Refractive surgery of any type within 1 year prior to screening in either eye.
20. Uncontrolled systemic disease of any type.
21. Anticipated alteration in chronic therapy with or introduction of agents known to have a substantial effect on IOP (e.g., alpha-adrenergic agonists, beta-adrenergic antagonists, calcium channel blockers, ACE inhibitors and/or angiotensin II receptor blockers), unless the subject and the medication dosage have been stable for three months prior to the screening visit and the dosage is not expected to change during the study.
22. Anticipated change in dosage of or introduction of new medications for chronic cardiac, pulmonary or hypertensive conditions.
23. Females who are pregnant or lactating and females of child-bearing potential who are not using a medically acceptable, highly effective method of birth control.
24. Current enrolment in an investigational drug or device study or participation in such a study within 30 days prior to screening.
25. History of drug or alcohol abuse.
26. Patient has any condition or situation that, in the Investigator's opinion, might confound the results of the study, may put the patient at significant risk or might interfere with the patient's ability to participate in the study.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sebastien Garrigue, PhD, Study Chair — Santen SAS
Locations (1):
- Hôpital des XV-XX, Paris, Île-de-France Region, France

RESULTS

PARTICIPANT FLOW:
Groups:
- DE-130A: DE-130A: Latanoprost 50 microg/ml preservative-free eye drops emulsion, eye drops emulsion in single-dose containers.
  Instillation of one drop, once daily in the evening (9 pm ±1 hour) in the conjunctival sac of the affected eye(s). Both eyes will be treated unless the patient suffers from unilateral OAG/OHT
- DE-130A/DE-130A: DE-130A: Latanoprost 50 microg/ml preservative-free eye drops emulsion, eye drops emulsion in single-dose containers.
  After 12 weeks, participants continued to use DE-130A for additional 12 months. Instillation of one drop, once daily in the evening (9 pm ±1 hour) in the conjunctival sac of the affected eye(s). Both eyes will be treated unless the patient suffers from unilateral OAG/OHT.
- Xalatan®/DE-130A: DE-130A: Latanoprost 50 microg/ml preservative-free eye drops emulsion, eye drops emulsion in single-dose containers.
  After 12 weeks, participants were converted to use DE-130A instead of Xalatan®. Instillation of one drop, once daily in the evening (9 pm ±1 hour) in the conjunctival sac of the affected eye(s). Both eyes will be treated unless the patient suffers from unilateral OAG/OHT.
Period: Period 1 Double Masked Treatment Period
Arm/Group | DE-130A | Xalatan® | DE-130A/DE-130A | Xalatan®/DE-130A
Started | 193 | 193 | 0 | 0
Completed | 190 | 190 | 0 | 0
Not Completed | 3 | 3 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Sponsor Temporarily Discontinued Study | 0 | 1 | 0 | 0
Period: Period 2 Open Label Treatment Period
Arm/Group | DE-130A | Xalatan® | DE-130A/DE-130A | Xalatan®/DE-130A
Started | 0 (After Double Masked Treatment Period 1, a sub-group of participants were moved to DE-130A/DE-130A Open Label Treatment Period 2.) | 0 (After Double Masked Treatment Period 1, a sub-group of participants were moved to DE-130A/DE-130A Open Label Treatment Period 2.) | 71 (After Double Masked Treatment Period, 71 participants from DE-130A Arm received DE-130A for additional 12 months in Open Label Treatment Period.) | 66 (After Double Masked Treatment Period, 66 participants from Xalatan Arm received DE-130A for additional 12 months in Open Label Treatment Period.)
Completed | 0 | 0 | 67 | 62
Not Completed | 0 | 0 | 4 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Early Termination | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DE-130A | Xalatan® | Total
Number analyzed (Participants) | 193 | 193 | 386
Age, Categorical [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description:
  Double Masked Period: 3-month treatment period, DE-130A vs Xalatan®: Randomization/baseline visit (Day 1), Week 4 (±3 days) and Week 12 (±3 days).
  Overall total number of baseline participants in the Double Masked Treatment Period are 384 subjects.
  Participants
    Double Masked Period: number analyzed (Participants) | 192 | 192 | 384
    Double Masked Period: <=18 years | 0 | 0 | 0
    Double Masked Period: Between 18 and 65 years | 102 | 94 | 196
    Double Masked Period: >=65 years | 90 | 98 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description:
  Double Masked Period: 3-month treatment period, DE-130A vs Xalatan®: Randomization/baseline visit (Day 1), Week 4 (±3 days) and Week 12 (±3 days).
  years
    Double Masked Period: number analyzed (Participants) | 192 | 192 | 384
    Double Masked Period | 62.3 (12.07) | 63.9 (10.14) | 63.1 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description:
  Double Masked Period: 3-month treatment period, DE-130A vs Xalatan®: Randomization/baseline visit (Day 1), Week 4 (±3 days) and Week 12 (±3 days).
  Participants
    Double Masked Period: number analyzed (Participants) | 192 | 192 | 384
    Double Masked Period: Female | 120 | 116 | 236
    Double Masked Period: Male | 72 | 76 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description:
  Double Masked Period: 3-month treatment period, DE-130A vs Xalatan®: Randomization/baseline visit (Day 1), Week 4 (±3 days) and Week 12 (±3 days).
  Participants
    Double Masked Period: number analyzed (Participants) | 192 | 192 | 384
    Double Masked Period: American Indian or Alaska Native | 0 | 0 | 0
    Double Masked Period: Asian | 4 | 4 | 8
    Double Masked Period: Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
    Double Masked Period: Black or African American | 0 | 0 | 0
    Double Masked Period: White | 184 | 186 | 370
    Double Masked Period: More than one race | 1 | 0 | 1
    Double Masked Period: Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Austria | 5 | 2 | 7
  Belgium | 5 | 6 | 11
  Estonia | 13 | 16 | 29
  Finland | 3 | 2 | 5
  France | 4 | 0 | 4
  Germany | 7 | 8 | 15
  Italy | 19 | 18 | 37
  Latvia | 14 | 12 | 26
  Poland | 4 | 5 | 9
  Spain | 19 | 24 | 43
  United Kingdom | 8 | 5 | 13
  Russia | 89 | 92 | 181
  South Korea | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) Change (mmHg) at Week 12
Description: Intraocular Pressure (IOP) change from baseline peak (mmHg). IOP was measured using calibrated Goldman applanation tonometer in the morning (9:00 am ± 1 hour). Analysis using Mixed-Effects Model for Repeated Measures (MMRM).
Time Frame: Week 12 (09:00) peak timepoint
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of the study medication and provided at least one post-baseline IOP measurement at peak and trough timepoints separately. The number analyzed are participants evaluable for the outcome measure at Week 12 (09:00) timepoint.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-130A | Xalatan®
Number analyzed (Participants) | 188 | 189
mmHg | -8.8 (0.25) | -8.2 (0.26)

2. Secondary Outcome: Corneal Fluorescein Staining (CFS) Change From Baseline (First Key Secondary Endpoint)
Description: CFS Change from baseline in participants with baseline CFS score ≥ 1 at Week 12
  Staining using fluorescein were graded using the Modified Oxford scale (7-point ordinal scale, score 0, 0.5, and 1 to 5 per area for cornea and conjunctiva separately) as shown below:
  * Score = 0: No staining dots
  * Score = 0.5: One staining dot per area
  * Score = 1: More staining dot per area than score 0.5
  * Score = 2: More staining dot per area than score 1
  * Score = 3: More staining dot per area than score 2
  * Score = 4: More staining dot per area than score 3
  * Score = 5: More staining dot per area than score 4
  A Mixed-Effects Model for Repeated Measures (MMRM) was fitted to the CFS change from baseline at each visit.
Time Frame: Week 12
Population: The number analyzed are participants evaluable for the outcome measure at Week 12 with CFS change from baseline in participants with baseline CFS score ≥ 1. Data were obtained by fitting a Mixed-Effects Model for Repeated Measures (MMRM) to the CFS change from baseline at each visit.
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | DE-130A | Xalatan®
Number analyzed (Participants) | 80 | 86
score | -0.71 (0.069) | -0.41 (0.077)

3. Secondary Outcome: Ocular Surface Disease (OSD) Symptoms (Average of 3 Symptoms); Second Key Secondary Endpoint
Description: Change from baseline in OSD symptom score (average of 3 symptoms: dry eye sensation, blurred/poor vision and burning/stinging/itching) in the study eye at Week 12 in patients with baseline symptom average score>0.
  Ocular symptoms were graded on a 5-point scale as shown below:
  * Scale = 0: Absent
  * Scale = 1: Mild
  * Scale = 2: Moderate
  * Scale = 3: Severe
  * Scale = 4: Very severe
  Least Square Means and p-values were obtained by fitting a Mixed-Effects Model for Repeated Measures (MMRM) model to the Ocular Surface Disease (OSD) average change from baseline at each visit.
Time Frame: Week 12
Population: The number analyzed are participants evaluable for the outcome measure at Week 12 with change from baseline in OSD symptom score>0 (average of 3 symptoms).
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | DE-130A | Xalatan®
Number analyzed (Participants) | 99 | 104
score | -0.26 (0.058) | -0.17 (0.060)

4. Primary Outcome: Intraocular Pressure (IOP) Change (mmHg) at Week 12
Description: Intraocular Pressure (IOP) change from baseline trough (mmHg). IOP was measured using calibrated Goldman applanation tonometer in the afternoon (4:00 pm ± 1 hour). Analysis using Mixed-Effects Model for Repeated Measures (MMRM).
Time Frame: Week 12 (16:00) trough timepoint
Population: Full Analysis Set (FAS) included all randomized subjects who received at least one dose of the study medication and provided at least one post-baseline IOP measurement at peak and trough timepoints separately. The number analyzed are participants evaluable for the outcome measure at Week 12 (16:00) timepoint.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | DE-130A | Xalatan®
Number analyzed (Participants) | 186 | 188
mmHg | -8.6 (0.24) | -8.1 (0.25)

ADVERSE EVENTS:
Time Frame: Period 1: 3-month from Randomization/baseline visit (Day 1), to Week 12 (±3 days). Period 2: 12-month follow-up from Week 12, from Week 12(±3 days) to Month 15 (± 1 week) visits. Adverse Events were collected from time of informed consent and were followed to resolution or until subject's participation in the study ended.
Description: Other Adverse Event data is a summary observed at a rate of 0% by System Organ Class and Preferred Term for both the Double Masked and Open Label Periods.
Arm/Group | DE-130A | Xalatan® | DE-130A/DE-130A | Xalatan®/DE-130A
All-Cause Mortality (participants affected / at risk) | 1/193 | 0/193 | 0/71 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/193 | 2/193 | 0/71 | 0/66
Other Adverse Events (participants affected / at risk) | 35/193 | 42/193 | 21/71 | 21/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE-130A (N=193) | Xalatan® (N=193) | DE-130A/DE-130A (N=71) | Xalatan®/DE-130A (N=66)
Acute Heart Failure (Cardiac disorders) | 1 | 0 | 0 | 0
Bilateral Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Patient Diagnosed With Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DE-130A (N=193) | Xalatan® (N=193) | DE-130A/DE-130A (N=71) | Xalatan®/DE-130A (N=66)
Ocular hyperaemia (Eye disorders) | 3 | 5 | 2 | 2
Conjunctival hyperaemia (Eye disorders) | 2 | 3 | 1 | 1
Dry eye (Eye disorders) | 2 | 1 | 1 | 0
Erythema of eyelid (Eye disorders) | 2 | 2 | 0 | 1
Keratitis (Eye disorders) | 2 | 0 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 0 | 2 | 1
Chalazion (Eye disorders) | 1 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 1 | 1 | 1
Eye pruritus (Eye disorders) | 1 | 3 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Growth of eyelashes (Eye disorders) | 1 | 0 | 2 | 2
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 1 | 2 | 1 | 2
Abnormal sensation in eye (Eye disorders) | 0 | 4 | 1 | 4
Eye irritation (Eye disorders) | 0 | 2 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 3 | 0 | 1
Lacrimal disorder (Eye disorders) | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Eye paraesthesia (Eye disorders) | 0 | 0 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 2 | 0 | 4
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Genital infection (Infections and infestations) | 0 | 1 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Burning mouth syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Instillation site pain (General disorders) | 0 | 3 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 2 | 0 | 0
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0
Dental implantation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT04133311/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT04133311/SAP_001.pdf